CLINICAL TRIAL: NCT06155617
Title: Development and Reliability of the PRESS to Function Approach: A Systematic Method for Upper Extremity Assessment
Brief Title: Pain, Range of Motion, Edema, Sensibility, Strength (PRESS) & Self-reported Function Create a Comprehensive Score
Acronym: PRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Howard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-20-PNAH-08
Record Dates: First submitted 2023-08-24; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-10

CONDITIONS: Hand Injuries and Disorders; Upper Extremity Problem
Keywords: PRESS to Function; Pain; Range of Motion; Edema; Sensation; Strength; Quick DASH; Upper Extremity; Hand
MeSH Terms: conditions — Hand Injuries; Disease; Pain; Edema

STUDY DESIGN:
Intervention Model Description: Single arm clinical trial. T-test employed to compare PRESS to Function scores before and after treatment. Reliability coefficient were computed to access consistency in the measurements of the Quick DASH and the PRESS to Function Scores
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Clinical Trial (Other): Participants with various upper extremity disorders are provided treatment/interventions and evaluated at baseline, 3-6 weeks, and at discharge using the PRESS to Function Approach
  Interventions: Other: Upper Extremity Rehabilitation

INTERVENTIONS:
Other: Upper Extremity Rehabilitation — Pain management, ROM, Edema Management, Desensitization, Strengthening, Functional Tasks

SUMMARY:
The aim of this study is to examine the development of a conceptual framework and provide evidence for reliability of a comprehensive hand therapy evaluation score. This approach provides a new standardized tool for upper extremity (UE) evaluation. Components of Pain, Range of Motion (ROM), Edema, Sensibility, Strength (PRESS), and self-reported Function were combined to create a baseline. Each assessment tool used for the PRESS to Function Approach assists in determining appropriate interventions.

DETAILED DESCRIPTION:
In this study, investigators used the innovative PRESS to Function Approach and Composite Score to describe the development and piloting of a systematic standard for upper extremity evaluation. Using existing instruments with substantial evidence of validity and reliability is more cost-effective than starting from scratch to develop and validate an instrument. This Approach and Score will provide occupational therapists an accurate measure to track the progression of a patient. The hypothesis for this study is Press to Function components will demonstrate utility for measuring clinical and patient-reported function when used as a comprehensive assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of upper extremity disorder as the primary diagnosis
* Surgical and nonsurgical Diagnoses
* Age 21 years or older

Exclusion Criteria:

* Concomitant Diseases (i.e cerebralvascular accident, cerebral palsy, spinal cord injury)
* Full Body Lymphedema
* Individuals who did not complete at least one reassessment

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Development and Reliability of PRESS to Function Approach: A Systematic Method for Upper Extremity Assessment | 4 weeks - 16 weeks depending on diagnosis and protocol
  The Development of the PRESS (pain, range of motion (ROM), edema, sensibility, strength) to Function Approach created a composite score. The PRESS to Function Composite Score combines subjective and objective measures to provide a single value to evaluate treatment prognosis. The six outcome measures (pain, ROM, edema, sensibility, strength, and function) were summed for 900 points to create a single score. The higher the score the less the overall disability.

SECONDARY OUTCOMES:
Pain Scale | 4 weeks - 16 weeks depending on diagnosis and protocol
  Pain was measured using the Numerical Pain Rating Scale (NPRS) and descriptors. The NPRS is indicative of a rating 0 through 10. The zero represents no pain and the 10 represents the worst imaginable pain
Range of Motion (ROM) | 4 weeks - 16 weeks depending on diagnosis and protocol
  For ROM, joints were measured with a goniometer. The unit of measurement is in degrees. Measurements range from 0 to 180 degrees. Each joint is compared to normative data. Zero represents the neutral and the least amount of motion.
Edema | 4 weeks - 16 weeks depending on diagnosis and protocol
  Edema considered both upper extremities (right and left) using a standard tape measure. The measurements were recorded according to units in centimeters (cm). Anatomical landmarks were chosen strategically for a ratio comparison as well as to establish baseline. Smaller numbers represent less edema or swelling.
Sensibility | 4 weeks - 16 weeks depending on diagnosis and protocol
  Sensibility was measured with Semmes Weinstein Monofilaments to determine sensory loss and touch pressure. The filaments are classified from grade 1 to 5 according to their thickness, where 5 represents the thinnest filament and 1 represents the largest filament: 1.65-2.83 = grade 5, 3.22-3.61 = grade 4, 3.84-4.31 = grade 3, 4.56-6.45 = grade 2, and 6.65 = grade 1
Strength (Grip and Pinch) | 4 weeks - 16 weeks depending on diagnosis and protocol
  Measured with the dynamometer and the pinch gauge in pounds. The higher the the number the stronger the patient. Strength may range from 0 pounds (weak) to 200 pounds (strong).There will be a comparison in some cases with normative data based on age and gender
Function with Quick Disability of the Arm, Shoulder, and Hand (DASH) | 4 weeks - 16 weeks depending on diagnosis and protocol
  The Quick DASH questionnaire is a Likert scale that uses 11 questions to measure the degree of difficulty in performing various physical activities. Due to a shoulder, arm, or hand problem questions address the severity of pain and tingling, the limitation on social activities, work, and sleep. All 11 self-report items must be completed to receive a score on a scale between 0-to-100 with the higher scores reflecting greater disability.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Ross, OTD, Principal Investigator — Howard University
Locations (1):
- Pinnacle Hand Therapy, Newport News, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Occupational Therapy Association. (2020). Occupational therapy practice framework: Domain and process (4th ed,) American Journal of Occupational Therapy, 74 ( Suppl. 2).
- [Result] Bohannon RW. Test-Retest Reliability of Measurements of Hand-Grip Strength Obtained by Dynamometry from Older Adults: A Systematic Review of Research in the PubMed Database. J Frailty Aging. 2017;6(2):83-87. doi: 10.14283/jfa.2017.8. PMID 28555708
- [Result] Hoe VC, Urquhart DM, Kelsall HL, Zamri EN, Sim MR. Ergonomic interventions for preventing work-related musculoskeletal disorders of the upper limb and neck among office workers. Cochrane Database Syst Rev. 2018 Oct 23;10(10):CD008570. doi: 10.1002/14651858.CD008570.pub3. PMID 30350850